CLINICAL TRIAL: NCT00885482
Title: Pilot Study for the Evaluation of the Safety and the Feasibility of Treatment Simplification to Atazanavir/Ritonavir + Lamivudine in Patients Stably Treated With Two NRTIs + Atazanavir/Ritonavir With Optimal Virologic Response.
Brief Title: Atazanavir and Lamivudine for Treatment Simplification
Acronym: AtLaS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Andrea De Luca, Professor, Catholic University of the Sacred Heart
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-011273-32
Record Dates: First submitted 2009-04-20; First posted 2009-04-22 (Estimated); Results first posted 2015-02-23 (Estimated); Last update posted 2015-03-13 (Estimated); Status verified 2015-02

CONDITIONS: HIV Infections
Keywords: HIV/AIDS; HAART; Simplification; Atazanavir; Lamivudine; treatment experienced
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Lamivudine; Atazanavir Sulfate; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm (Experimental): Treatment simplification from a "standard" combined antiretroviral therapy including 2 NRTIs and Atazanavir with Ritonavir to Lamivudine plus Atazanavir with Ritonavir. Treatment simplification from three-drugs- to two-drugs-based antiretroviral therapy.
  Interventions: Drug: Lamiduvine (Epivir); Drug: Atazanavir (Reyataz); Drug: Ritonavir (Norvir)

INTERVENTIONS:
Drug: Lamiduvine (Epivir) — Epivir 300 mg
Drug: Atazanavir (Reyataz) — Reyataz 300 mg
Drug: Ritonavir (Norvir) — Norvir 100 mg

SUMMARY:
Objectives of the study:

1. To verify the safety of the study treatment, defined as the persistent control of the virus' replication at 48 weeks after the simplification to lamivudine + atazanavir with ritonavir.
2. To collect relevant information about the safety and the metabolic impact of this strategy in order to eventually design a non-inferiority randomized controlled trial for the evaluation of the safety and the efficacy of this strategy in the future.

DETAILED DESCRIPTION:
Combined antiretroviral therapy has greatly improved the natural history of HIV infection/AIDS. Yet, it is associated with important short- and long- term side effects. In particular, nucleoside and nucleotide analogs may cause anemia, pancreatitis, mitochondrial dysfunction, lactic acidosis, lipoatrophy and reduction of renal function or of bone density.

Our study aims to verify the safety and efficacy of a simplification of a dual therapy (Lamivudine plus Atazanavir with Ritonavir), confiding on the potency and high genetic barrier of ritonavir-boosted agents.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with the same regimen including 2NRTIs + ATV/r from at least 6 months
* Aged 18 years or older
* Who gave informed consent to the participation to the study
* With at least two viral load < 50 copies/mL in two consecutive determinations at least 3 months apart
* With CD4 cell count > 200 cells/μL and absence of any opportunistic infection or AIDS-related disease by one year at least

Exclusion Criteria:

* Pregnancy or breast feeding, desire of pregnancy in the short term
* Previous virological failure to antiretroviral therapy and/or previous exposure to mono- or dual therapies with reverse transcriptase nucleosidic analogues
* Patients with insufficient atazanavir plasma through concentration (lower than 0.23 μg/mL at 12th hour or 0.15 μg/mL at 24th hour) at screening and/or at baseline
* Patients with grade 3 or 4 laboratory abnormalities at screening (except for glucose or lipid serum levels and direct or indirect bilirubin)
* Concomitant treatment with antacids or proton-pump blockers or any other drug with known interactions or contraindications with the study medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-05; Primary Completion 2010-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea De Luca, MD, Principal Investigator — Catholic University of Sacred Heart
Locations (1):
- Catholic University of Sacred Heart, Rome, Italy

REFERENCES:
- [Derived] Fabbiani M, Bracciale L, Doino M, D'Avino A, Marzocchetti A, Navarra P, Cauda R, De Luca A, Di Giambenedetto S. Tenofovir discontinuation could predispose to urolithiasis in atazanavir-treated patients. J Infect. 2011 Apr;62(4):319-21. doi: 10.1016/j.jinf.2011.02.004. Epub 2011 Feb 15. No abstract available. PMID 21329725

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Arm
Started | 40
Completed | 36
Not Completed | 4
Not completed — Pregnancy | 1
Not completed — Lack of Efficacy | 1
Not completed — Death | 1
Not completed — low Therapeutic drug monitoring (TDM) | 1

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 38
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 23
Region of Enrollment [Number; unit: participants]
  Italy | 40

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Virological Failure (Two Consecutive Measures of HIV-RNA Higher Than 50 Copies/mL or a Single Measure Higher Than 1000 Copies/mL) Within 48 Weeks at intention-to.Treat Analysis
Time Frame: 48 weeks
Measure: Number; unit: patients
Arm/Group | Single Arm
Number analyzed (Participants) | 40
patients | 1

2. Secondary Outcome: Time to Virological Failure at Survival Analysis
Time Frame: 48 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Number of Patients With Viral Load Lower Than 50 Copies/mL at 48 Weeks at the Intention to Treat Analysis
Time Frame: 48 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Evolution of CD4 Cell Count During the 48 Weeks
Time Frame: 48 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Evolution of Adherence and Quality of Life During the 48 Weeks
Time Frame: 48 weeks
Reporting Status: Not Posted

6. Secondary Outcome: Evolution of Atazanavir Plasma Concentrations During the 48 Weeks
Time Frame: 48 weeks
Reporting Status: Not Posted

7. Secondary Outcome: Change of Metabolic Parameters at 48 Weeks
Time Frame: 48 weeks
Reporting Status: Not Posted

8. Secondary Outcome: Change of the Results of Neurocognitive Tests at 48 Weeks
Time Frame: 48 weeks
Reporting Status: Not Posted

9. Secondary Outcome: Change of Bone Density and of Subcutaneous Fat at 48 Weeks
Time Frame: 48 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Single Arm
Serious Adverse Events (participants affected / at risk) | 6/40
Other Adverse Events (participants affected / at risk) | 15/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm (N=40)
renal colics (Renal and urinary disorders) | 4 (4)
hypertensive crisis (Vascular disorders) | 1 (1)
brain hemorrage and subsequent myocardial infarction (Cardiac disorders) | 1 (2) — Brain hemorrage ans subsequent death for myocardial infarction in a 63 years old female, with a previous history of head trauma and hypertension; events not judged as drug-related since they happened in a high-risk patient
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm (N=40)
fever (Infections and infestations) | 15 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes